CLINICAL TRIAL: NCT04085991
Title: Two TraCer PositROn EmiSSion Tomography ComBination for Efficacy EstimatiOn of Prostate Specific Membrane Antigen Radioligand Therapy in Patients With Metastatic Prostate Cancer
Acronym: CROSSBOW
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug no longer available
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, MD, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROSSBOW
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostatic Neoplasms; Metastatic Prostate Cancer; Metastatic Prostatic Adenocarcinoma; Metastatic Prostate Carcinoma in the Soft Tissue
Keywords: Radioligand therapy; PSMA; PSMA therapy; 1095
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 131I-PSMA-1095 Radioligand Therapy (RLT) (Experimental): Intravenous injection of 100 mCi of 131I-PSMA-1095 RLT, Q8 weeks up to a maximum of 4 doses
  Interventions: Drug: 131I-PSMA-1095 Radioligand Therapy (RLT)

INTERVENTIONS:
Drug: 131I-PSMA-1095 Radioligand Therapy (RLT) — Intravenous injection of 100 mCi of 131I-PSMA-1095, Q8 weeks up to a maximum of 4 doses.
  Other Names: PSMA RLT

SUMMARY:
Single-arm, open-label, phase II trial in 200 competent adult male patients with Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-3 and progressive metastatic prostate cancer, failing, failed, refused, not eligible for or no access to further approved lines of therapy. Patients will undergo sequential FDG positron emission tomography (PET) and 18F-DCFPyL PET to assess FDG/DCFPyL concordance fraction. Patients with DCFPyL/FDG concordance of 50% or greater will be treated with 131I-PSMA-1095 radioligand therapy (RLT). Best post-treatment serum prostate specific antigen response will be compared to concordance fraction.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18 years or older
* Documented metastatic adenocarcinoma of the prostate
* Under active medical oncology care
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Able to tolerate the physical requirements of two PET/CT scans including lying for up to 30 minutes
* Progressive disease on any of: bone scan, CT, MRI or serum PSA as judged by the investigator
* Serum prostate specific antigen ≥ 1 ng/ml at baseline or CT/MRI soft-tissue measurable disease as per RECIST v1.1
* Failed, failing, refused, no access to or not eligible for any approved prostate cancer therapies including but not limited to: ADT, NAAD (e.g., abiraterone, enzalutamide, darolutamide or apalutamide), docetaxel, cabazitaxel, radium-223 and oligometastatic RTX
* Life expectancy of at least 3 months as judged by the investigator

Exclusion Criteria:

* Medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Exceeding the weight limit of the PET/CT bed (approximately 400 lbs.) or who cannot fit through the PET/CT bore (approximately 70 cm diameter)
* Unmanageable claustrophobia
* Prior failure of PSMA RLT
* Prior hemi-body irradiation
* Impaired organ function as evidenced by any of the following laboratory values:

  * Absolute neutrophil count < 1.5 x109/L
  * Platelet count < 75 x109/L
  * Hemoglobin < 85 g/L
  * Albumin < 2.5 g/dL (25 g/L)
  * Total bilirubin > 2 x ULN (unless in instances of Gilbert's disease)
  * AST or ALT > 2.5 x ULN (or > 5.0 x ULN in the presence of liver metastases)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only.
Enrollment: 11 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Serum prostate specific antigen (PSA) | 3 months post last dose of RLT
  The best serum prostate specific antigen (PSA) response will be calculated for each patient as: pre-treatment PSA minus lowest post-treatment PSA divided by pre-treatment PSA. Best PSA response will be reported as percent reduction (or increase) from baseline.

SECONDARY OUTCOMES:
Adverse events | 3 months post last dose of RLT
  Frequency of adverse events in participants receiving therapy as per CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Probst, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Stephan Probst, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No